CLINICAL TRIAL: NCT01202435
Title: An Open-Label, Multiple-Dose, Randomized, 2-Way Crossover Study In Healthy Volunteers To Determine The Steady-State Pharmacokinetics Of The 82.5 Mg Pregabalin Controlled Release Formulation Administered Following An Evening Meal Relative To The 25 Mg Of The Immediate Release Formulation Administered Three Times Daily
Brief Title: An Investigation Of The Absorption And Pharmacokinetics Of Multiple Doses Of A Controlled Release Pregabalin Tablet As Compared To Multiple Doses Of The Immediate Release Pregabalin Capsule
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A0081215
Record Dates: First submitted 2010-09-14; First posted 2010-09-15 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2010-12

CONDITIONS: Healthy
Keywords: pregabalin; pharmacokinetics; bioavailability; bioequivalence
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregabalin controlled release, 82.5 mg (Experimental)
  Interventions: Drug: Pregabalin controlled release, 82.5 mg
- Pregabalin immediate release, 25 mg (Other): Reference Treatment
  Interventions: Drug: Pregabalin immediate release, 25 mg

INTERVENTIONS:
Drug: Pregabalin controlled release, 82.5 mg — 82.5 mg controlled release tablet administered once daily for four days.
  Arms: Pregabalin controlled release, 82.5 mg
Drug: Pregabalin immediate release, 25 mg — 25 mg immediate release capsules administered three times daily for four days
  Arms: Pregabalin immediate release, 25 mg

SUMMARY:
The purpose of this study is to 1)evaluate the extent of absorption of multiple doses of a pregabalin controlled release tablet as compared to multiple doses of the pregabalin immediate release capsule, 2) evaluate the pharmacokinetics of multiple doses of a pregabalin controlled release tablet as compared to multiple doses of pregabalin immediate release capsule and 3) evaluate the safety and tolerability of multiple doses of a pregabalin controlled release tablet as compared to multiple doses of the pregabalin immediate release capsule.

DETAILED DESCRIPTION:
Evaluate the absorption, pharmacokinetics, safety/tolerability of multiple doses of a pregabalin controlled release tablet as compared to multiple doses of pregabalin immediate release capsule

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or females
* Between the ages of 18 and 55 years, inclusive
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2

Exclusion Criteria:

* Illicit drug use
* Pregnant or nursing females
* Females of childbearing potential who are unwilling or unable to use an acceptable method of contraception

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Area under the curve at steady-state over a 24 hour period (AUC24)for assessment of equivalence between 82.5 mg CR and 25 mg IR capsule given 3 times daily (total daily dose 75 mg) | 5 days

SECONDARY OUTCOMES:
Safety endpoints include evaluation of adverse events | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- [Derived] Chew ML, Alvey CW, Plotka A, Pitman VW, Alebic-Kolbah T, Scavone JM, Bockbrader HN. Pregabalin controlled-release pharmacokinetics in healthy volunteers: analysis of four multiple-dose randomized clinical pharmacology studies. Clin Drug Investig. 2014 Sep;34(9):627-37. doi: 10.1007/s40261-014-0221-2. PMID 25078977
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081215&StudyName=An%20Investigation%20Of%20The%20Absorption%20And%20Pharmacokinetics%20Of%20Multiple%20Doses%20Of%20A%20Controlled%20Release%20Pregabalin%20Tablet%20As%20Compared%20To%20Multi